CLINICAL TRIAL: NCT03273387
Title: The Role of Trimetazidine on Right Ventricle Function in Pulmonary Arterial Hypertension Patients in National Cardiovascular Center Harapan Kita Hospital Indonesia
Brief Title: The Role of Trimetazidine on Right Ventricle Function in Pulmonary Arterial Hypertension
Acronym: TRIMETA-PH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Hary Sakti Muliawan, MD, PhD, MD,PhD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LB.02.01/VII/172/KEP.009/2017
Record Dates: First submitted 2017-09-03; First posted 2017-09-06 (Actual); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Precapillary Pulmonary Hypertension
MeSH Terms: interventions — Trimetazidine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugar pill (Placebo Comparator): The participant will received placebo oral capsule bid for 3 months on top of their regular PAH specific therapy.
  Interventions: Drug: Placebo oral capsule
- trimetazidine (Experimental): The participant will received trimetazidine 35 mg bid for 3 months on top of their regular PAH specific therapy.
  Interventions: Drug: Trimetazidine

INTERVENTIONS:
Drug: Trimetazidine — The participant will received trimetazidine 35 mg bid for 3 months on top of their regular PAH specific therapy.
  Other Names: Trizedon MR
  Arms: trimetazidine
Drug: Placebo oral capsule — The participant will received placebo oral capsule bid for 3 months on top of their regular PAH specific therapy.
  Other Names: sugar pill
  Arms: Sugar pill

SUMMARY:
The study will evaluate the effect of trimetazidine versus placebo in addition to standard pulmonary arterial hypertension regime on right ventricular function in pulmonary arterial hypertension patients.

DETAILED DESCRIPTION:
Right ventricular dysfunction is the worst mortality predictor in pulmonary arterial hypertension (PAH). Recent study has described that approximately 25% of PAH patients will developed into right ventricular failure despite therapeutic reduction of pulmonary vascular resistance. Subsequently, several studies have shown that fatty acid accumulation in right ventricle was inversely correlated with right ventricular function in PAH patients. Several PAH animal studies have revealed that metabolic glucose oxidation impairment through increased aerobic glycolysis, mitochondrial dysfunction, and lipotoxicity play significant role in right ventricular failure. Moreover, several pulmonary hypertension animal studies have demonstrated the benefit of partial fatty acid inhibitor such as trimetazidine on right ventricle function. It was hypothesize that trimetazidine improved right ventricular function through indirect effect of increased glucose oxidation by blocking the Randle cycle. Therefore, we hypothesize that trimetazidine can improve right ventricular function in pulmonary arterial hypertension patients.

ELIGIBILITY:
Inclusion Criteria:

* Pre-capillary Pulmonary Hypertension patients assessed by right heart catheterization
* Signed informed consent

Exclusion Criteria:

* Patient belonging to post-capillary, Isolated post-capillary, or combined post -capillary and pre-capillary pulmonary hypertension according to 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension.
* Moderate to severe chronic pulmonary obstructive disease
* Right Ventricular Ejection Fraction > 45% assessed by cardiac magnetic resonance.
* Documented left ventricular dysfunction with left ventricular ejection fraction < 50% assessed by cardiac magnetic resonance.
* Severe renal impairment (Serum creatinine > 2.5 mg/dL, eGFR < 30ml/min/1.73 m^2, or routine dialysis treatment).
* Malignant arrhythmia such as total atrioventricular block or ventricular fibrillation or unstable ventricular tachycardia.
* Patients who are receiving or have been receiving any investigational drugs within 1 month before the baseline visit
* Acute or chronic impairment (other than dyspnea) limiting the ability to comply with study requirements
* Psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements
* Females who are lactating or pregnant or those who plan to become pregnant during the study
* Known Parkinson disease
* Known hypersensitivity to any of the drug formulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hary Sakti Muliawan, MD,PhD, Principal Investigator — Department Cardiology and Vascular Medicine Universitas Indonesia
Locations (1):
- National Cardiovascular Center Harapan Kita Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from NCCHK PH outpatient clinic from September 2017 until November 2018
Pre-assignment Details: A total of 35 Patients were enrolled between September 2017 and November 2018 at NCCHK PAH outpatient clinic. A total of 26 patients were consent to underwent the trial and randomly assigned to receive trimetazidine or placebo with ratio 1:1.
Period: Overall Study
Arm/Group | Sugar Pill | Trimetazidine
Started | 13 | 13
Completed | 10 | 10
Not Completed | 3 | 3
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Trimetazidine | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (3.8) | 48 (1.5) | 48 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Percentage of gender differences in our PAH patients.
  Participants
    Female | 11 | 12 | 23
    Male | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13 | 13 | 26
onset of diagnosis to study [Mean (Standard Deviation); unit: days] — The number of days since first diagnosed with PAH until intervention. The longer the onset of diagnosis to study intervention suggest longer the patients suffered from PAH which may or may not correlated with PAH severity
  days | 1170 (387) | 926 (214) | 1048 (1093)
SF-36 Functional Capacity [Mean (Standard Deviation); unit: units on a scale] — SF-36 functional capacity score is an questionnaire instrument which evaluate quality of life including functional capacity. The SF-36 functional capacity score scale from 0-100 with better functional capacity along with higher scale.
  units on a scale | 61.15 (4.77) | 46.54 (5.44) | 53.84 (19.56)
WHO Functional Class [Count of Participants; unit: Participants] — Percentage of participant with WHO functional class II or III on each group. WHO functional class II defines as PAH patients with slight limitation of physical activity. They are comfortable at rest. Ordinary activity causes dyspnea, fatigue, chest pain, or syncope.
  WHO functional class III defines as PAH patients with marked limitation of physical activity. They are comfortable with rest. Less than ordinary activities causes dyspnea, fatigue, chest pain or syncope.
  Participants
    WHO functional class II | 9 | 4 | 13
    WHO functional class III | 4 | 9 | 13
Glomerular Filtration Rate [Mean (Standard Deviation); unit: ml/min/1.73 m^2] | 96.6 (7.9) | 110.7 (3.9) | 106 (15.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.3 (3.8) | 21 (0.8) | 22.1 (8.6)
Phosphodiesterase-5 inhibitor [Count of Participants; unit: Participants] — Percentage of participant with Phosphodiesterase-5 inhibitor treatment.
  Participants | 12 | 12 | 24
Prostacyclin analogue (beraprost) [Count of Participants; unit: Participants] — Percentage of participants with oral prostacyclin analogue (beraprost) treatment
  Participants | 8 | 5 | 13
beta blocker [Count of Participants; unit: Participants] — Percentage of participant with beta blocker treatment.
  Participants | 5 | 8 | 13
ACE-inhibitor [Count of Participants; unit: Participants] — Percentage of participant with ACE-Inhibitor treatment.
  Participants | 4 | 5 | 9
Angiotensin receptor II blocker [Count of Participants; unit: Participants] — Percentage of participant with Angiotensin receptor II blocker treatment.
  Participants | 4 | 1 | 5
Warfarin [Count of Participants; unit: Participants] — Percentage of participant with warfarin treatment.
  Participants | 4 | 6 | 10
spironolactone [Count of Participants; unit: Participants] — Percentage of participant with spironolactone treatment.
  Participants | 9 | 10 | 19
furosemide [Count of Participants; unit: Participants] — Percentage of participant with furosemide treatment.
  Participants | 11 | 8 | 19
digoxin [Count of Participants; unit: Participants] — Percentage of participant with digoxin treatment.
  Participants | 1 | 2 | 3
mean Right atrial pressure [Mean (Standard Deviation); unit: mmHg] | 5.9 (1.4) | 6 (1.2) | 5.9 (3.9)
mean pulmonary arterial pressure [Mean (Standard Deviation); unit: mmHg] | 62 (5.9) | 59 (3.6) | 60 (11.2)
LV end diastolic pressure [Mean (Standard Deviation); unit: mmHg] | 7.2 (1.2) | 7.8 (0.8) | 7.4 (3.1)
RV end diastolic volume [Mean (Standard Deviation); unit: ml] | 258 (28) | 260 (31) | 259 (83)
RV end systolic volume [Mean (Standard Deviation); unit: ml] | 193 (20) | 206 (25) | 197 (67)
RV ejection fraction [Mean (Standard Deviation); unit: %] | 24.5 (2.8) | 21.1 (4.4) | 22.4 (10)
LV end diastolic volume [Mean (Standard Deviation); unit: ml] | 79 (6.3) | 83 (5.3) | 81 (18)
LV end systolic volume [Mean (Standard Deviation); unit: ml] | 29 (2.8) | 33 (3.3) | 31 (9.7)
LV ejection fraction [Mean (Standard Deviation); unit: %] | 64 (2.6) | 59 (2.4) | 62 (7.5)
Native T1 anteroseptal [Mean (Standard Deviation); unit: ms] — Native T1 is measuring the T1 tissue using CMR with MOLLI technique at 1.5 T which normal value ranged between 900 to 1100ms.
  Native T1 is increased in edema, inflammation, cellular edema, myocyte necrosis, and fibrosis.
  ms | 993 (612) | 1354 (441) | 1164 (555)
Native T1 septal [Mean (Standard Deviation); unit: ms] | 1108 (512) | 1110 (411) | 1109 (454)
Native T1 inferoseptal [Mean (Standard Deviation); unit: ms] | 930 (418) | 1474 (736) | 1187 (637)
Native T1 Lateral [Mean (Standard Deviation); unit: ms] | 1090 (470) | 1357 (473) | 1216 (478)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Right Ventricular Ejection Fraction (RVEF %) After 3 Months Intervention
Description: Right ventricular ejection fraction (RVEF %) assessed by Cardiac MRI at 3 months intervention minus with RVEF at baseline.
Time Frame: Baseline and 3 months after intervention
Population: A total 13 patients were assigned to each group equally. There were 6 patients who were not able to complete the study. A total of 2 patients from both group died due to RV failure. One patients from trimetazidine group withdrawn due to atypical angina and one patients from placebo group withdrawn due to claustrophobia.
Measure: Mean (Standard Error); unit: percentage of ejected blood
Arm/Group | Sugar Pill | Trimetazidine
Number analyzed (Participants) | 10 | 10
percentage of ejected blood | -2.8 (1.6) | 3.9 (1.5)
Statistical Analysis 1: Comparison: Sugar Pill vs Trimetazidine; Test type: Superiority; p = 0.008, t-test, 2 sided — 95% Confidence interval 1.97 - 11.3 statistical significant if p<0.05; t=2.988 df=18

2. Secondary Outcome: Changes in Cardiac Fibrosis After 3 Months Intervention
Description: Native T1 mapping (ms) assessed by Cardiac MRI at 3 months intervention minus with Native T1 at baseline.
Time Frame: Baseline and 3 months after intervention
Measure: Mean (Standard Error); unit: ms
Arm/Group | Sugar Pill | Trimetazidine
Number analyzed (Participants) | 10 | 10
ms
  Native T1 anteroseptal | 138 (555) | 190 (538)
  Native T1 Septal | 292 (677) | 371 (670)
  Native T1 Inferoseptal | 294 (618) | -123 (645)
  Native T1 Lateral | 287 (744) | -194 (487)
Statistical Analysis 1: Comparison: Sugar Pill vs Trimetazidine; Test type: Superiority; p = 0.33, two-way ANOVA — statistical significant if p <0.05; DF=3

3. Secondary Outcome: Changes in Functional Capacity After 3 Month Intervention
Description: Functional capacity assessed by SF-36 score after 3 month intervention minus with functional capacity at baseline.
  SF-36 functional capacity score scale 0 to 100 with better functional capacity along with higher score.
Time Frame: Baseline and 3 months after intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sugar Pill | Trimetazidine
Number analyzed (Participants) | 10 | 10
score on a scale | -17.73 (3.72) | 11.5 (5.27)
Statistical Analysis 1: Comparison: Sugar Pill vs Trimetazidine; Test type: Superiority; p = 0.0002, t-test, 2 sided — 95% Confidence interval 15.92 to 42.53 statistical significant if p <0.05; t=4.598 df=19

ADVERSE EVENTS:
Time Frame: three months for each intervention.
Description: safety population included all participants who received at least one dose of intervention.
Arm/Group | Sugar Pill | Trimetazidine
All-Cause Mortality (participants affected / at risk) | 2/13 | 2/13
Serious Adverse Events (participants affected / at risk) | 2/13 | 2/13
Other Adverse Events (participants affected / at risk) | 1/13 | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=13) | Trimetazidine (N=13)
Cardiovascular mortality (Cardiac disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=13) | Trimetazidine (N=13)
paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
musculoskeletal angina (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT03273387/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT03273387/ICF_001.pdf